CLINICAL TRIAL: NCT01853839
Title: Treatment Adherence to JNC 7(Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure, 7th Report) Guidelines in Cardiovascular (CV)-Risk Patients Across the Middle East - the Impact of Ramadan Fasting on Achieving Treatment Goals in Daily Practice
Brief Title: Impact of Ramadan on Achieving Joint National Committee (JNC) 7 Treatment Goals in CV Risk Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.602
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This is an out-patient based prospective, multi-centre, observational post-marketing surveillance study amongst internists and cardiologists. In this study, patients with essential hypertension and at least one additional risk factor will be included. Patients may take any antihypertensive treatment which is approved for cardiovascular protection including Micardis 80 mg / Micardis Plus. Patients will be followed over one year in four visits from baseline to endpoint with an additional visit before and after the month of Ramadan.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Male or female of age 18 years or older;
2. Newly diagnosed and untreated or previously treated and uncontrolled patients with essential hypertension;
3. Seated blood pressure of >140/90 mmHg or >130/80 mmHg in patients with diabetes mellitus or chronic kidney disease;
4. Patients with at least one cardiovascular (cv) risk factor;
5. Ability to provide written informed consent.

Exclusion criteria:

1. Patients with contraindications to the prescribed antihypertensive medications;
2. Pregnant or lactating women or women of childbearing potential not using an acceptable method of contraception;
3. Patients who are participating in any other study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients wih at least one CV risk factor
Sampling Method: Non-Probability Sample
Enrollment: 1674 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (132):
- Algeria (26):
  - Boehringer Ingelheim Investigational Site 106, Algiers
  - Boehringer Ingelheim Investigational Site 107, Algiers
  - Boehringer Ingelheim Investigational Site 108, Algiers
  - Boehringer Ingelheim Investigational Site 109, Algiers
  - Boehringer Ingelheim Investigational Site 110, Algiers
  - Boehringer Ingelheim Investigational Site 111, Algiers
  - Boehringer Ingelheim Investigational Site 112, Algiers
  - Boehringer Ingelheim Investigational Site 113, Algiers
  - Boehringer Ingelheim Investigational Site 114, Algiers
  - Boehringer Ingelheim Investigational Site 115, Algiers
  - Boehringer Ingelheim Investigational Site 116, Algiers
  - Boehringer Ingelheim Investigational Site 117, Algiers
  - Boehringer Ingelheim Investigational Site 118, Algiers
  - Boehringer Ingelheim Investigational Site 119, Algiers
  - Boehringer Ingelheim Investigational Site 120, Algiers
  - Boehringer Ingelheim Investigational Site 121, Algiers
  - Boehringer Ingelheim Investigational Site 122, Algiers
  - Boehringer Ingelheim Investigational Site 123, Algiers
  - Boehringer Ingelheim Investigational Site 124, Algiers
  - Boehringer Ingelheim Investigational Site 125, Algiers
  - Boehringer Ingelheim Investigational Site 126, Algiers
  - Boehringer Ingelheim Investigational Site 127, Algiers
  - Boehringer Ingelheim Investigational Site 128, Algiers
  - Boehringer Ingelheim Investigational Site 129, Algiers
  - Boehringer Ingelheim Investigational Site 130, Algiers
  - Boehringer Ingelheim Investigational Site 131, Algiers
- Egypt (31):
  - Boehringer Ingelheim Investigational Site 29, Al Fayyum
  - Boehringer Ingelheim Investigational Site 15, Alexandria
  - Boehringer Ingelheim Investigational Site 19, Alexandria
  - Boehringer Ingelheim Investigational Site 21, Alexandria
  - Boehringer Ingelheim Investigational Site 22, Alexandria
  - Boehringer Ingelheim Investigational Site 23, Alexandria
  - Boehringer Ingelheim Investigational Site 3, Alexandria
  - Boehringer Ingelheim Investigational Site 6, Alexandria
  - Boehringer Ingelheim Investigational Site 18, Asyut
  - Boehringer Ingelheim Investigational Site 27, Asyut
  - Boehringer Ingelheim Investigational Site 11, Banisuif
  - Boehringer Ingelheim Investigational Site 10, Cairo
  - Boehringer Ingelheim Investigational Site 12, Cairo
  - Boehringer Ingelheim Investigational Site 13, Cairo
  - Boehringer Ingelheim Investigational Site 14, Cairo
  - Boehringer Ingelheim Investigational Site 17, Cairo
  - Boehringer Ingelheim Investigational Site 1, Cairo
  - Boehringer Ingelheim Investigational Site 20, Cairo
  - Boehringer Ingelheim Investigational Site 24, Cairo
  - Boehringer Ingelheim Investigational Site 25, Cairo
  - Boehringer Ingelheim Investigational Site 26, Cairo
  - Boehringer Ingelheim Investigational Site 28, Cairo
  - Boehringer Ingelheim Investigational Site 2, Cairo
  - Boehringer Ingelheim Investigational Site 4, Cairo
  - Boehringer Ingelheim Investigational Site 5, Cairo
  - Boehringer Ingelheim Investigational Site 7, Cairo
  - Boehringer Ingelheim Investigational Site 8, Cairo
  - Boehringer Ingelheim Investigational Site 9, Cairo
  - Boehringer Ingelheim Investigational Site 30, Domiat
  - Boehringer Ingelheim Investigational Site 16, Menia
  - Boehringer Ingelheim Investigational Site 31, Tanta
- Lebanon (29):
  - Boehringer Ingelheim Investigational Site 66, Beirut
  - Boehringer Ingelheim Investigational Site 67, Beirut
  - Boehringer Ingelheim Investigational Site 68, Beirut
  - Boehringer Ingelheim Investigational Site 69, Beirut
  - Boehringer Ingelheim Investigational Site 70, Beirut
  - Boehringer Ingelheim Investigational Site 71, Beirut
  - Boehringer Ingelheim Investigational Site 72, Beirut
  - Boehringer Ingelheim Investigational Site 73, Beirut
  - Boehringer Ingelheim Investigational Site 74, Beirut
  - Boehringer Ingelheim Investigational Site 75, Beirut
  - Boehringer Ingelheim Investigational Site 76, Beirut
  - Boehringer Ingelheim Investigational Site 77, Beirut
  - Boehringer Ingelheim Investigational Site 78, Beirut
  - Boehringer Ingelheim Investigational Site 79, Beirut
  - Boehringer Ingelheim Investigational Site 80, Beirut
  - Boehringer Ingelheim Investigational Site 81, Beirut
  - Boehringer Ingelheim Investigational Site 82, Beirut
  - Boehringer Ingelheim Investigational Site 83, Beirut
  - Boehringer Ingelheim Investigational Site 84, Beirut
  - Boehringer Ingelheim Investigational Site 85, Beirut
  - Boehringer Ingelheim Investigational Site 86, Beirut
  - Boehringer Ingelheim Investigational Site 87, Beirut
  - Boehringer Ingelheim Investigational Site 88, Tripoli
  - Boehringer Ingelheim Investigational Site 89, Tripoli
  - Boehringer Ingelheim Investigational Site 90, Tripoli
  - Boehringer Ingelheim Investigational Site 91, Tripoli
  - Boehringer Ingelheim Investigational Site 92, Tripoli
  - Boehringer Ingelheim Investigational Site 93, Tripoli
  - Boehringer Ingelheim Investigational Site 94, Tripoli
- Saudi Arabia (35):
  - Boehringer Ingelheim Investigational Site 35, Dammam
  - Boehringer Ingelheim Investigational Site 36, Dammam
  - Boehringer Ingelheim Investigational Site 37, Dammam
  - Boehringer Ingelheim Investigational Site 38, Hofuf
  - Boehringer Ingelheim Investigational Site 50, Jeddah
  - Boehringer Ingelheim Investigational Site 51, Jeddah
  - Boehringer Ingelheim Investigational Site 52, Jeddah
  - Boehringer Ingelheim Investigational Site 53, Jeddah
  - Boehringer Ingelheim Investigational Site 54, Jeddah
  - Boehringer Ingelheim Investigational Site 55, Jeddah
  - Boehringer Ingelheim Investigational Site 56, Jeddah
  - Boehringer Ingelheim Investigational Site 57, Jeddah
  - Boehringer Ingelheim Investigational Site 58, Jeddah
  - Boehringer Ingelheim Investigational Site 59, Jeddah
  - Boehringer Ingelheim Investigational Site 60, Jeddah
  - Boehringer Ingelheim Investigational Site 61, Jeddah
  - Boehringer Ingelheim Investigational Site 62, Jeddah
  - Boehringer Ingelheim Investigational Site 63, Jeddah
  - Boehringer Ingelheim Investigational Site 64, Jeddah
  - Boehringer Ingelheim Investigational Site 65, Jeddah
  - Boehringer Ingelheim Investigational Site 32, Khobar
  - Boehringer Ingelheim Investigational Site 33, Khobar
  - Boehringer Ingelheim Investigational Site 34, Khobar
  - Boehringer Ingelheim Investigational Site 105, Riyadh
  - Boehringer Ingelheim Investigational Site 39, Riyadh
  - Boehringer Ingelheim Investigational Site 40, Riyadh
  - Boehringer Ingelheim Investigational Site 41, Riyadh
  - Boehringer Ingelheim Investigational Site 42, Riyadh
  - Boehringer Ingelheim Investigational Site 43, Riyadh
  - Boehringer Ingelheim Investigational Site 44, Riyadh
  - Boehringer Ingelheim Investigational Site 45, Riyadh
  - Boehringer Ingelheim Investigational Site 46, Riyadh
  - Boehringer Ingelheim Investigational Site 47, Riyadh
  - Boehringer Ingelheim Investigational Site 48, Riyadh
  - Boehringer Ingelheim Investigational Site 49, Riyadh
- United Arab Emirates (11):
  - Boehringer Ingelheim Investigational Site 100, Dubai
  - Boehringer Ingelheim Investigational Site 101, Dubai
  - Boehringer Ingelheim Investigational Site 102, Dubai
  - Boehringer Ingelheim Investigational Site 103, Dubai
  - Boehringer Ingelheim Investigational Site 104, Dubai
  - Boehringer Ingelheim Investigational Site 132, Dubai
  - Boehringer Ingelheim Investigational Site 95, Sharjah city
  - Boehringer Ingelheim Investigational Site 96, Sharjah city
  - Boehringer Ingelheim Investigational Site 97, Sharjah city
  - Boehringer Ingelheim Investigational Site 98, Sharjah city
  - Boehringer Ingelheim Investigational Site 99, Sharjah city

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients are included a non-completers if they did not meet the definition of the intention-to-treat (ITT) population (all patients, who received at least one dose of study medication) or if the subject attended the week 52 visit less than 26 weeks after baseline.
Groups:
- All Subjects: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  All antihypertensive drugs will be prescribed and administered according to the approved prescribing information in the country where the patient resides. Treatment duration is up to 52 weeks.
Period: Overall Study
Arm/Group | All Subjects
Started | 2092
Completed | 1663
Not Completed | 429
Not completed — Violated inclusion criteria | 2
Not completed — Not meet ITT population definition | 58
Not completed — End of treatment visit too early | 33
Not completed — Lost to follow-up or no valid BP measure | 336

BASELINE CHARACTERISTICS:
Population: All subjects included in the study according to the study protocol i.e. patients who did not violate any inclusion or exclusion criteria
Arm/Group | All Subjects
Number analyzed (Participants) | 2090
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information was only collected for 1979 participants.
  years | 54.78 (11.01)
Gender [Number; unit: participants] — Gender information was only collected for 1969 participants.
  participants
    Female | 808
    Male | 1161

OUTCOME MEASURES:

1. Primary Outcome: Achievement of the JNC 7 Treatment Goals (BP <140/90 mmHg) at Week 52
Description: The proportion of patients enrolled in the study who achieve the JNC 7 (the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure) treatment goals (blood pressure (BP) <140/90 mmHg) in a primary-care setting at week 52. This variable was derived from the mean sitting blood pressure assessed by the investigators at week 52. To achieve JNC 7 treatment goals, the subject had to satisfy both blood pressure criteria - systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg.
Time Frame: Up to 52 weeks
Population: ITT dataset which included all patients, who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Groups:
- All Subjects: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  Treatment duration is up to 52 weeks.
Arm/Group | All Subjects
Number analyzed (Participants) | 1663
Percentage of participants
  Yes | 94.95
  No | 5.05

2. Secondary Outcome: Achieving JNC 7 Treatment Goals After Ramadan
Description: The proportion of patients enrolled in the study who achieve the JNC 7 (the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure) treatment goals (blood pressure (BP) <140/90 mmHg) in a primary-care setting after Ramadan. This variable was derived from the mean sitting blood pressure assessed by the investigators after Ramadan. To achieve JNC 7 treatment goals, the subject had to satisfy both blood pressure criteria - systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg.
Time Frame: 1 month
Population: Per-protocol (PP) population which included all eligible patients who did not experience any protocol violation and were treated with the study medication up to week 52 (study completers) according to the prescribing information.
Measure: Number; unit: Percentage of participants
Groups:
- Fasting: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  Treatment duration is up to 52 weeks. Patients who did fast for Ramadan.
- Non-Fasting: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  Treatment duration is up to 52 weeks. Patients who did not fast for Ramadan.
Arm/Group | Fasting | Non-Fasting
Number analyzed (Participants) | 1230 | 164
Percentage of participants
  Yes | 87.07 | 85.97
  No | 12.93 | 14.02

3. Secondary Outcome: Cardiovascular Events
Description: Percentage of participants who experienced a major cardiovascular (CV) event
Time Frame: Up to 52 weeks
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 2090
Percentage of participants | 0.91

4. Secondary Outcome: The Overall Assessment of Treatment by Patients at 52 Weeks
Description: The overall assessment of treatment by patients at 52 weeks. Assessed using a verbal rating scale with 5 categories: Outstanding, very satisfactory, satisfactory, marginal and not satisfactory.
Time Frame: Up to 52 weeks
Population: Per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1548
Percentage of participants
  Outstanding | 25.45
  Very satisfactory | 53.88
  Satisfactory | 18.80
  Marginal | 1.42
  Not satisfactory | 0.45

5. Secondary Outcome: The Overall Assessment of Treatment by Physicians at 52 Weeks
Description: The overall assessment of treatment by physicians at 52 weeks. Assessed using a verbal rating scale with 5 categories: Outstanding, very satisfactory, satisfactory, marginal and not satisfactory.
Time Frame: Up to 52 weeks
Population: Per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1548
Percentage of participants
  Outstanding | 25.97
  Very satisfactory | 55.49
  Satisfactory | 16.21
  Marginal | 1.74
  Not satisfactory | 0.58

6. Secondary Outcome: Compliance of Patients up to 10 Days Before Ramadan
Description: Compliance of patients up to 10 days before ramadan (treated by internists and cardiologists as primary physician). Subjects were asked how often they have not taken their medicine and were given five possible choices from "none of the time" to "all of the time".
Time Frame: 10 days before Ramadan
Population: Per-protocol population including all patients with data 10 days before Ramadan
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1788
Percentage of participants
  None of the time | 70.58
  Some of the time | 25.45
  Most of the time | 0.95
  All the time | 1.06
  Do not know | 1.96

7. Secondary Outcome: Compliance of Patients up to 10 Days After Ramadan
Description: Compliance of patients up to 10 days after Ramadan (treated by internists and cardiologists as primary physician). Subjects were asked how often they have not taken their medicine and were given five possible choices from "none of the time" to "all of the time".
Time Frame: 10 days after Ramadan
Population: Per-protocol population including all patients with data 10 days after Ramadan
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1748
Percentage of participants
  None of the time | 71.11
  Some of the time | 24.37
  Most of the time | 2.40
  All the time | 0.80
  Do not know | 1.32

8. Secondary Outcome: Compliance of Patients During the Whole Study Duration (52 Weeks)
Description: Compliance of patients during the whole study duration (treated by internists and cardiologists as primary physician). Subjects were asked how often they have not taken their medicine and were given five possible choices from "none of the time" to "all of the time".
Time Frame: Up to 52 weeks
Population: Per-protocol population including all patients with data at 52 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1668
Percentage of participants
  None of the time | 70.68
  Some of the time | 25.78
  Most of the time | 1.98
  All the time | 0.48
  Do not know | 1.08

9. Secondary Outcome: Achievement of the JNC 7 Treatment Goals During the Whole Study Duration (Treated by Internists and Cardiologists as Primary Physician)
Description: Proportion of patients who achieved the JNC 7 treatment goals during the whole study duration (treated by internists and cardiologists as primary physician)
Time Frame: Up to 52 weeks
Population: Per-protocol population
Measure: Number; unit: Percentage of participants
Groups:
- Cardiologist: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  Treatment duration is up to 52 weeks. Patients whose primary physician was a cardiologist.
- Internist: Newly diagnosed or uncontrolled adult hypertensive patients with at least one cardiovascular risk factor who are prescribed antihypertensive drugs with an approved indication for cardiovascular protection (including Micardis® 80 mg/ Micardis® Plus tablets) as monotherapy or as part of a combination regimen with other antihypertensive agents.
  Treatment duration is up to 52 weeks. Patients whose primary physician was a internist.
Arm/Group | Cardiologist | Internist
Number analyzed (Participants) | 864 | 382
Percentage of participants
  Yes | 96.64 | 93.98
  No | 3.36 | 6.02

10. Secondary Outcome: The Difference in Systolic Blood Pressure Before and After the Month of Ramadan
Description: Change from baseline in systolic blood pressure before and after the month of Ramadan
Time Frame: Baseline, 10 days before Ramadan, 10 days after Ramadan and 52 weeks
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fasting | Non-Fasting
Number analyzed (Participants) | 1210 | 160
mmHg
  10 days before Ramadan (N=1200, 153) | 24.4 (16.7) | 25.0 (16.3)
  10 days after Ramadan (N=1190, 160) | 28.3 (17.0) | 29.3 (15.0)
  52 weeks (N=1210, 160) | 30.3 (17.2) | 30.6 (15.9)

11. Secondary Outcome: The Difference in Diastolic Blood Pressure Before and After the Month of Ramadan
Description: Change from baseline in diastolic blood pressure before and after the month of Ramadan
Time Frame: Baseline, 10 days before Ramadan, 10 days after Ramadan and 52 weeks
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fasting | Non-Fasting
Number analyzed (Participants) | 1210 | 160
mmHg
  10 days before Ramadan (N=1200, 153) | 12.2 (9.6) | 12.5 (10.4)
  10 days after Ramadan (N=1190, 160) | 14.4 (9.6) | 15.1 (9.2)
  52 weeks (N=1210, 160) | 15.5 (9.9) | 16.2 (10.2)

12. Secondary Outcome: The Percentage of Patients Achieving JNC 7 Treatment Goals at the End of the 1 Year Treatment Duration
Description: The proportion of patients enrolled in the study who achieve the JNC 7 (the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure) treatment goals (blood pressure (BP) <140/90 mmHg) in a primary-care setting at the end of the 1 year treatment duration. This variable was derived from the mean sitting blood pressure assessed by the investigators at the end of the 1 year treatment duration. To achieve JNC 7 treatment goals, the subject had to satisfy both blood pressure criteria - systolic blood pressure below 140 mm Hg and diastolic blood pressure below 90 mm Hg. At this timepoint, a diagnosis of diabetes mellitus and/or kidney disease was also taken into account. Subjects with either of the mentioned conditions had to have systolic blood pressure lower than 130 mm Hg and diastolic blood pressure below 80 mm Hg to satisfy JNC 7 treatment goals.
Time Frame: Up to 52 weeks
Population: Per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1578
Percentage of participants
  Yes | 85.93
  No | 14.07

13. Secondary Outcome: Adverse Events Under Angiotensin II (Type 1) Receptor Blockers (ARBs) Treatment When Given in Combination With Calcium-Channel Blockers (CCBs)
Description: Number of participants with adverse events in participants receiving Angiotensin II (Type 1) Receptor Blockers (ARBs) when given in combination with Calcium-Channel Blockers (CCBs) during the whole study duration.
Time Frame: Up to 52 weeks
Population: All subjects who took a combination of ARB and CCB drugs.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 518
participants | 27

ADVERSE EVENTS:
Time Frame: From drug administration until end of study, 52 weeks
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 21/2090
Other Adverse Events (participants affected / at risk) | 0/2090
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=2090)
Acute myocardial infarction (Cardiac disorders) | 17
Accidental death (General disorders) | 1
Sudden death (General disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.